CLINICAL TRIAL: NCT05553925
Title: Implementation of an Online Weight Management Program in Clinical and Community Settings
Brief Title: Partnerships for Reducing Overweight and Obesity with Patient-Centered Strategies 2.0
Acronym: PROPS2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Heather J. Baer, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000605
Record Dates: First submitted 2022-08-18; First posted 2022-09-26 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: The investigators will implement the combined intervention (online weight management program plus coaching and patient navigator support) as part of standard of care for at least 5,000 patients with overweight or obesity. All eligible patients, in each participating Brigham and Women's Hospital practice/site, who wish to enroll will receive the intervention. The investigators will invite a sample of enrolled patients to participate in a single-arm, longitudinal study to assess changes in patient-reported outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Implementation (Experimental): At least 5,000 patients from the participating BWH practices/sites will receive the combined intervention (online weight management program with patient navigator support and personalized coaching) as part of standard of care for overweight and obesity.
  Interventions: Other: Online Weight Management Program with Coaching and Patient Navigator Support

INTERVENTIONS:
Other: Online Weight Management Program with Coaching and Patient Navigator Support — Patients will enroll in a 12-month digital health program available in online and mobile versions with live, personalized coaching and patient navigator support.
  Patient Interface
  * Digital scale and Fitbit
  * Brief lessons that focus on helping patients improve their nutrition, exercise, sleep, and stress
  * Weight, diet, and physical activity tracking
  * Regular, personalized feedback and support from a health coach
  * Spanish Version
  Patient navigators are non-licensed staff. Their responsibilities will include enrolling patients in the program, monitoring their progress, and updating providers periodically. They also will be able to connect patients with additional resources and services, such as the Center for Weight Management and Wellness, if appropriate.

SUMMARY:
The primary objective of the project is to adapt and implement a combined weight management intervention (an online program plus coaching and patient navigator support) across multiple settings and a diverse cross-section of patients and providers affiliated with Brigham and Women's Hospital (BWH).

The overall goals of the proposed project are:

1. To improve management of overweight and obesity in clinical and community settings.
2. To improve outcomes among patients with overweight or obesity.

To accomplish these goals, the investigators will engage with various stakeholders to adapt the combined intervention, implement the intervention across multiple settings and a diverse cross-section of patients and providers affiliated with BWH, evaluate the impact of the implementation, and create an implementation guide for dissemination.

The specific aims of the proposed project are as follows:

Aim 1: To continue to engage with patients, providers, and other stakeholders to adapt and integrate the intervention in a variety of clinical and community settings.

Aim 2: To implement the intervention in a variety of patients and settings and to evaluate its impact on outcomes, using the RE-AIM framework.

Aim 3: To evaluate maintenance of the intervention six months after formal implementation activities have ended, and to prepare a detailed implementation guide to help increase future reach and uptake.

DETAILED DESCRIPTION:
The investigators will recruit patients and providers from the following practices/sites affiliated with Brigham and Women's Hospital. Other sites may be included, if appropriate:

* BWH Primary Care Center of Excellence
* Division of Cardiovascular Medicine at BWH Heart & Vascular Center
* BWH Division of Endocrinology, Diabetes, and Hypertension
* BWH Department of Orthopedic Surgery
* BWH Comprehensive Breast Health Center (only B-PREP program)
* BWH Center for Community Wellness at Sportsman's Tennis & Enrichment Center
* BWH Center for Weight Management and Wellness
* BWH Nutrition and Wellness Service (within the Department of Nutrition)
* BWH Division of Sleep and Circadian Disorders

Pre- and Post-Implementation Focus Groups, Interviews, and Surveys:

The investigators will conduct focus groups and/or semi-structured interviews with approximately 15-20 patients, before and after implementing the intervention, to understand their attitudes and experiences with weight management and to obtain feedback on their thoughts about the proposed intervention. Patients will be eligible for the focus groups and interviews if they are receiving medical care at one of the participating BWH practices/sites, are over 20 years old, and have a BMI of 25 kg/m2 or higher. In addition, patients must speak English to participate in the focus groups and interviews.

The investigators will recruit 15-20 providers from the participating clinics for voluntary, semi-structured interviews and administer a survey to all providers in the clinics before and after implementing the intervention. Providers may include staff physicians, residents or fellows, nurse practitioners or physician assistants, and additional staff who provide services to patients, including dietitians and patient navigators. The goal will be to evaluate their views and practices around management of overweight and obesity, obtain feedback about the proposed intervention workflow, and identify any other barriers or facilitators to implementing the intervention. Providers will be eligible to participate if they practice in one of the participating BWH clinics.

Intervention Implementation:

The investigators will enroll at least 5,000 eligible patients from across the participating BWH practices/sites. The intervention will be offered as standard of care to all eligible patients at participating BWH practices/sites. Eligible patients will be enrolled in the program for 12 months. After patients register for the online program, they will complete lessons about nutrition, physical activity, sleep, and stress; track their diet, physical activity, and weight; and interact with a coach, who will provide personalized feedback and support. Patient navigators also will monitor patients' progress, periodically update providers, and help refer/connect them to other resources for weight management, if appropriate. The investigators will invite a sample of 300-500 patients who are enrolled in the intervention to complete an online survey at the beginning and end of their enrollment. The goal will be to assess changes in patient-reported outcomes, such as diet, physical activity, and health status.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 years or over
2. Have a healthcare provider at BWH (received care from a primary care provider or specialist at BWH in last 24 months)
3. Have a primary care provider
4. BMI of 30 or over OR
5. BMI 25 to 29.9 kg/m2 plus ≥ 1 with indicators for increased cardiovascular risk or other obesity-related comorbidity (e.g., type 2 diabetes, prediabetes, high blood pressure, hyperlipidemia, sleep apnea, non-alcoholic fatty liver disease)
6. English- or Spanish-speaking
7. Regular Internet access (at least once per week) via smartphone, computer, or tablet and valid email address (required to register for the online program)

Exclusion Criteria:

1. Patients who are pregnant
2. Patients who have Type 1 diabetes OR on insulin for treatment of diabetes
3. Patients receiving comfort care measures, hospice, or nursing home
4. Patients with a serious medical condition for which weight loss is contraindicated (e.g., end stage renal disease, active cancer (other than non-melanoma skin cancer)
5. Patients who have had bariatric or endoscopic surgery in last 12 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
Weight Change | Baseline and 12 months
  Weight change over 12 months, calculated from patients' weights recorded from digital scales, manually entered in the online program, and/or recorded in the electronic health record at visits. These weights will be used to calculate weight change over 12 months among enrolled patients and the number/proportion of enrolled patients who achieve ≥ 5% weight loss over 12 months.

SECONDARY OUTCOMES:
Reach | Every month for 14 months
  The number, proportion, and description of end-users receiving the intervention, including the number of patients who are referred by their provider, who are identified via the electronic health record, or who self-refer to the program. Data from the electronic health record and other internal databases will be used to track the total number and proportion of patients who are referred or identified, as well as the number and proportion who are screened, eligible, enrolled, and registered for the program.
Patient Satisfaction | 12 months after enrollment in the program
  Patient satisfaction with the intervention as self-reported by patients on surveys and during interviews. Data also will identify barriers and facilitators.
Diet | Baseline and 12 months
  Changes in patients' diet during the 12-month intervention, as self-reported on surveys.
Physical Activity | Baseline and 12 months
  Changes in patients' physical activity during the 12-month intervention, as self-reported on surveys.
Health Status | Baseline and 12 months
  Changes in patients' health status during the 12-month intervention, as self-reported on surveys.
Self-efficacy Around Weight Loss | Baseline and 12 months
  Changes in patients' self-efficacy around weight loss during the 12-month intervention, as self-reported on surveys.
Change in hemoglobin A1c (HbA1c) | Baseline and 12 months
  Changes in Hb1Ac over 12 months (only among patients with type 2 diabetes). This will be calculated from HbA1c values recorded in the electronic health record.
Changes in Blood Pressure | Baseline and 12 months
  Changes in systolic and diastolic blood pressure over 12 months. This will be calculated from blood pressure values recorded in the electronic health record.
Engagement with the Online Program | During 12 months of enrollment in the program
  Engagement with the online program will be measured by the number/proportion of enrolled patients who engage with each of the following components of the online program: log meals, text and/or call coach, log sleep, log weight, complete an activity, complete a lesson. Data will be retrieved from the vendor database.
Weight Change at 18 Months | 18 Months (six months after program completion)
  Weight change at 18 months. This will be calculated from weight values recorded in the patients' electronic health records and will be used to evaluate whether patients maintained weight lost at 12 months (primary outcome) at 18 months, six months after they complete the online program.

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Baer, Sc.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No